CLINICAL TRIAL: NCT03497637
Title: Comparison of Non-Invasive Vessel Fractional Flow Reserve Calculated From Angiographic Images Versus Fractional Flow Reserve in Patients With Intermediate Coronary Artery Stenoses
Brief Title: Comparison of Vessel-FFR Versus FFR in Intermediate Coronary Stenoses
Acronym: LIPSIASTRATEGY
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Helios Health Institute GmbH (Other)
Collaborators: Heart Center Leipzig - University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HRC045277
Record Dates: First submitted 2018-04-06; First posted 2018-04-13 (Actual); Last update posted 2024-11-25 (Actual); Status verified 2024-11

CONDITIONS: Coronary Artery Disease; Coronary Artery Stenoses
MeSH Terms: conditions — Coronary Artery Disease; Coronary Stenosis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pd/Pa guided Therapy (Active Comparator): use of resting distal coronary pressure to aortic pressure ratio (Pd/Pa) to assess the hemodynamic significance of coronary stenoses
  Interventions: Diagnostic Test: measurement of Pd/Pa
- FFR guided therapy (Active Comparator): use of pressure-derived FFR to assess the hemodynamic significance of coronary stenoses
  Interventions: Diagnostic Test: measurement of FFR

INTERVENTIONS:
Diagnostic Test: measurement of FFR — use of pressure-derived FFR to assess the hemodynamic significance of coronary stenoses
  Arms: FFR guided therapy
Diagnostic Test: measurement of Pd/Pa — use of resting distal coronary pressure to aortic pressure ratio (Pd/Pa) to assess the hemodynamic significance of coronary stenoses
  Arms: Pd/Pa guided Therapy

SUMMARY:
This is a prospective, randomized, controlled, multicenter, open-label study designed to assess whether vFFR is non-inferior to FFR in assessment of intermediate coronary stenosis in terms of the occurrence of MACE during 12 months after randomization.

DETAILED DESCRIPTION:
Coronary angiography is insensitive to assess the physiologic significance of a coronary stenosis. Therefore, clinical guidelines support the use of pressure-derived fractional flow reserve (FFR) to assess the hemodynamic significance of coronary stenosis. Nevertheless, the penetration of FFR in clinical routine continues to be limited by its requirement for pharmacological vasodilation, prolonged procedure time and adverse systemic effects from adenosine.

Vessel-FFR (vFFR) is a novel method for evaluating the functional significance of coronary stenosis by calculation of the pressure drop in the vessel based on computation of two angiographic projections. The vFFR values at each point along the vessel are color-coded and superimposed on the 3D epicardial model and cut-off values of ≤0.80 identical to standard invasive FFR apply.

These developments may translate towards more physiology guided intervention bearing the potential to improve clinical outcomes in patients with stable CAD. The ability to derive FFR values from routinely performed coronary angiograms, without the practical drawbacks that limit invasive techniques, could have an important impact on daily clinical practice.

To date no randomized outcome-based clinical trial has compared an image-based FFR methodology with standard invasive FFR in terms of subsequent clinical outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years
* Willing to participate and able to understand, read and sign the informed consent document before the planned procedure
* Eligible for coronary angiography and/or PCI
* Coronary artery disease in one or more native major epicardial vessels or their branches by coronary angiogram with visually assessed de novo coronary stenosis in which the physiological severity of the lesion is in question (typically 40-80% diameter stenosis).
* Stable angina or acute coronary syndrome (non-culprit vessels only and outside of primary intervention during acute STEMI or NSTE-ACS)
* Participation in another interventional study

Exclusion Criteria:

* Previous CABG with patent grafts to the interrogated vessel
* Tandem stenoses separated by more than 10 mm that require separate pressure guide wire interrogation or PCI (not to be interrogated or treated as a single stenosis)
* Total coronary occlusions
* Hemodynamic instability (Killip class III-IV)
* Heavily calcified or tortuous vessels
* Terminal disease with life expectancy of less than 12 months
* STEMI within 48 hours of procedure
* Severe valvular heart disease
* ACS patients with difficulty in assessing which the culprit lesion is
* Significant contraindication to adenosine administration (e.g. Asthma bronchiale)
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1054 (Estimated)
Dates: Start 2020-10-23 (Actual); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-11-01 (Estimated)

PRIMARY OUTCOMES:
Major Adverse Cardiac Event (MACE) rate | 1 year
  composite of cardiac death, non-fatal myocardial infarction or unplanned revascularization

SECONDARY OUTCOMES:
MACE during long-term follow-up | 2 and 5 years
Each component of the primary endpoint assessed by structured telephone interview and verification by hospital reports | 1, 2 and 5 years
Repeat revascularization (PCI or CABG) assessed by structured telephone interview and verification by hospital reports in case of event | 1, 2 and 5 years
All-cause mortality | 1, 2 and 5 years
Cross-over rate from the one strategy to the other | at intervention
Number of analyzable lesions in both treatment arms | at intervention

CONTACTS AND LOCATIONS:
Overall Officials: Holger Thiele, MD, Principal Investigator — Heart Center Leipzig - University Hospital
Locations (8):
- Germany (8):
  - Heart Center Dresden - University Clinic, Dresden
  - University Clinic Erlangen, Erlangen
  - Universitätsklinikum Essen, Essen
  - University Clinic Giessen and Marburg, Giessen
  - Herzzentrum Leipzig, Leipzig
  - University Clinic Leipzig, Leipzig
  - Klinikum der Stadt Ludwigshafen, Ludwigshafen
  - Lukaskrankenhaus Neuss, Neuss

IPD SHARING:
Plan to Share IPD: No